CLINICAL TRIAL: NCT00801307
Title: A Single Site,Exploratory,Phase I/II,Randomised Trial Comparing the Effect of He/O2 Mixtures(He/O2 78:22 and He/O2 65:35) to Medical Air on Pulmonary Function in Moderate/Severe Asthma and COPD Patients and Healthy Volunteers
Brief Title: Trial Comparing Effect of He/O2 to Medical Air on Pulmonary Function Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Air Liquide SA (Industry)
Collaborators: Inamed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ALMED-07-C2-012; 2007-004158-10 (EudraCT Number)
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; Healthy
Keywords: evaluate Inspiratory Capacity (IC) measured by spirometry
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): He/O2 78:22
  Interventions: Device: spirometer
- 2 (Experimental): He/O2 65:35
  Interventions: Device: spirometer
- 3 (Active Comparator): Medical Air
  Interventions: Device: spirometer

INTERVENTIONS:
Device: spirometer — According to the randomisation order, the appropriate medical gas cylinder with the pressure regulator will be connected to a humidifier to avoid the inhalation of very dry gas; the humidifier will be connected to the breathing bag; the flow of the medical gas will be adjusted individually for each subject/patient by the valve of the pressure regulator.
  Other Names: ergospirometer

SUMMARY:
This clinical trial will include healthy volunteers, COPD patients and asthmatic patients who will breathe He/O2 78:22, He/O2 65:35 and medical air consecutively in a randomised order.

DETAILED DESCRIPTION:
Two types of measurements will be performed with each of the three evaluated gases:

* pulmonary function measurements at rest to establish the resistance to airflow in a reproducible way, including the measurements of Inspiratory Capacity (IC), Forced Expiratory Volume in 1 second (FEV1), Forced Expiratory Flows (FEF) at different lung volumes (25 to 75% of the vital capacity), and Forced Vital Capacity (FVC),
* Tidal Volume (TV) measured at rest and during light cycling exercise. The results of this study should be useful to evaluate the extent of influence on gas concentration, since none of the previous trials have been performed with He/O2 65:35, as well as the extent of influence on the lung disease, since none of the previous trials have been performed with asthmatic patients at various disease stages.

The working hypothesis is that when using He/O2 mixtures 78:22 and 65:35, the flow resistance decreases as compared to medical air because low density helium replaces nitrogen, thus resulting in a lower workload of breathing for asthmatic and COPD patients. For patients with reduced pulmonary function, this difference might result in greater Inspiratory Capacity.

That is why Inspiratory Capacity will be measured as primary efficacy criterion, but also Tidal Volume and other pulmonary function parameters on 3 types of subjects/patients :

* healthy volunteers,
* patients with moderate and severe persistent asthma,
* patients with moderate and severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* All subjects/patients:

  * Willing and able to complete the requirements of this study including the signature of the written informed consent,
  * Able to complete the study in 5 working days or less,
  * Able to perform pulmonary function tests
* Healthy volunteers:

  * Never smoker or subject who stopped smoking at least 6 months before selection (strictly less than 10 pack-years),
  * Having pulmonary function tests within the normal range(according to predicted values for age, sex and height as referenced in ATS/ERS 1993 standards)
* Patients with moderate/severe persistent asthma:

  * Documented clinical diagnosis of moderate or severe persistent asthma (according to GINA 2006 guidelines),
  * Stable asthma in the 4 weeks prior to selection as evidenced by no change in asthma medication, no treatment for asthma in an emergency,acute care setting and no admission to hospital for acute asthma

Patients with moderate / severe COPD:

* Aged ≥ 45 and £ 80 years old,
* Documented clinical diagnosis of moderate or severe COPD(according to GOLD 2006 guidelines),
* With a smoking history of 10 pack-years or more,
* Stable COPD in the 4 weeks prior to selection as evidenced by no change in COPD medication, no treatment for COPD in an emergency, acute care setting and no admission to hospital for COPD exacerbation

Exclusion Criteria:

* Obese subject/patient having a Body Mass Index (BMI) > 35,
* Past or present respiratory disease including being free from the common cold and rhinitis for at least 4 weeks before selection except asthma for asthmatic patients and COPD for COPD patients,
* Daily need for 12 hours or more of long term oxygen therapy,
* Pregnant or lactating woman,
* Lack of efficient contraception according to CPMP/ICH 286/95 note 31,
* Any contra-indication to perform pulmonary function tests or light cycling exercise,
* Clinically significant or uncontrolled pathologic conditions which may interfere with the study procedures,
* Drug abuse or psychic disorders resulting in an inability to fully understand the requirements of the study,
* Legal status which prohibits informed consent,
* Participation in any interventional clinical trial within 30 days prior to selection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Inspiratory Capacity measured by spirometry at rest while breathing each He/O2 mixture compared to its measurement on medical air | 30 mn

SECONDARY OUTCOMES:
Inspiratory Capacity measured by ergospirometry while breathing Pulmonary function parameters at rest, i.e., FEV1, FVC, FEF25-75, PEF and ERV while breathing each He/O2 mixture compared to medical air, | 20 Mn

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, Dr. med., Principal Investigator — Inamed Research GmbH & Co. KG
Locations (1):
- Inamed Research GmbH & Co. KG, Robert-Koch-Allee 2, Gauting, Germany